CLINICAL TRIAL: NCT02763501
Title: Comparing a Randomised Controlled Intervention With Observational Data.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Region Örebro County (Other)
Collaborators: The Scandinavian Obesity Surgery Registry (Unknown)
Responsible Party: Principal Investigator, Erik Stenberg, MD, DR, Region Örebro County
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EPN 2015/097
Record Dates: First submitted 2016-05-03; First posted 2016-05-05 (Estimated); Last update posted 2016-10-17 (Estimated); Status verified 2016-10

CONDITIONS: Obesity, Morbid
Keywords: bariatric surgery; gastric bypass; intestinal obstruction; postoperative complication; methods; laparoscopy
MeSH Terms: conditions — Obesity, Morbid; Intestinal Obstruction; Postoperative Complications

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- RCT (Active Comparator): patients operated with laparoscopic gastric bypass surgery within a register based RCT from May 1st 2010 until Nov 14th 2011.
  1:1 randomization to closure of mesenteric defects by running, non-absorbable sutures
  Interventions: Procedure: closure of mesenteric defects; Procedure: non-closure of mesenteric defects
- non-RCT (Active Comparator): patients operated with laparoscopic gastric bypass surgery outside of the RCT from May 1st 2010 until Nov 14th 2011.
  Intervention of mesenteric defects according to local tradition or choice of surgeon (non-randomized)
  Interventions: Procedure: closure of mesenteric defects; Procedure: non-closure of mesenteric defects

INTERVENTIONS:
Procedure: closure of mesenteric defects — Closure of mesenteric defects by use of non-absorbable running sutures in RCT; and according to the choice of the surgeon in the non-RCT
Procedure: non-closure of mesenteric defects — Mesenteric defects are left open

SUMMARY:
Comparison of participants in a randomised controlled trial (RCT) with observational data from patients operated in Sweden during the same period of time. The primary objective is to compare effects from a complex surgical intervention from RCT and observational data.

DETAILED DESCRIPTION:
Randomised controlled trials (RCT) are "golden standard" for assessing interventions in medical science. Due to ethical or practical reasons, RCTs may however not always be feasible. The study objective was to test if the results from the RCT differ from observational data in a setting with a complex surgical intervention.

Using the Scandinavian Obesity Surgery Registry database we intend to compare patients operated with laparoscopic gastric bypass surgery within a register based RCT from May 1st 2010 until Nov 14th 2011, with all patients operated with the same procedure registered in the database during the same period of time.

Primary end-point measures are severe complications within 30 days (safety outcome) and surgery for small bowel obstruction (efficacy outcome) within 4 years.

ELIGIBILITY:
Inclusion Criteria:

* The same as acceptance criteria for bariatric surgery according to the 1991 NIH Consensus Statement

Exclusion Criteria:

* retrocolic gastric bypass procedure
* previous bariatric procedures
* primary open procedures
* missing data on handling of the mesenteric defects

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10992 (Actual)
Dates: Start 2010-05; Primary Completion 2014-12 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
severe postoperative complications within 30 days | 30 days
  Specified as Clavien-Dindo grade 3b or more
reoperation for small bowel obstruction | 4 years
  Efficacy outcome: Number of participants with reoperation due to small bowel obstruction defined as acute symptoms of bowel obstruction with findings suggestive of small bowel obstruction during surgery

SECONDARY OUTCOMES:
postoperative length of stay | 30 days
length of the operation | intraoperative
specific postoperative complications | 30 days
  leakage or deep intra-abdominal infection, bleeding requiring intervention, small bowel obstruction/ileus, port-related complications, wound dehiscence, other wound complications (mainly superficial wound infections), anastomotic stricture, marginal ulcer, cardiovascular length of the operation event, pulmonary complication (other than pulmonary embolism), venous thromboembolism (including pulmonary embolism), urinary tract infection and other (in this case specified) complication
weight-loss at 2 years after surgery | 2 years
  specified as excessive weight-loss (% excess weight loss = 100 x [initial weight-postoperative weight]/[initial weight-weight corresponding to BMI 25 kg/m2])

IPD SHARING:
Plan to Share IPD: No
Group data will be published. Deidentified individual participant data for all primary and secondary outcomes will be available after study completion.

REFERENCES:
- See also: The Scandinavian Obesity Surgery Registry — http://www.ucr.uu.se/soreg